CLINICAL TRIAL: NCT05944887
Title: Does Intravenous Lidocaine Reduce Propofol Consumption and the Side Effects of Sedation During Gastroscopy in ASA 1 and 2 Patients.
Brief Title: Intravenous Lidocaine to Reduce Propofol Consumption During Gastroscopy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Omar Assam, principal investigator, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: P2023/236
Record Dates: First submitted 2023-06-19; First posted 2023-07-13 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Diagnostic Gastroscopy
MeSH Terms: interventions — Lidocaine; Propofol; Gastroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: computered randomisation, sealed enveloppes linisol versus placebo prepared by anesthesist not involved in the study or in patient care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Linisol (Active Comparator): Patients will receive 1.5 mg/kg of intravenous linisol before propofol sedatation and gastroscope introduction
  Interventions: Drug: Lidocaine 2% Injectable Solution; Drug: Propofol injection; Procedure: gastroscopy
- Sham (Placebo Comparator): Patients will receive intravenous placebo (saline solution),before propofol sedation and gastroscope introduction
  Interventions: Drug: Saline administration as placebo; Drug: Propofol injection; Procedure: gastroscopy

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — administration of a bolus of lidocaine 1.5 mg/kg
  Arms: Linisol
Drug: Saline administration as placebo — administration of a bolus of saline solution as a placebo
  Arms: Sham
Drug: Propofol injection — Sedation by total intravenous administration (TIVA) of propofol
Procedure: gastroscopy — esogastroduodenoscopy

SUMMARY:
The goal of this clinical trial is to assess if intravenous administration of linisol reduce the propofol consumption and the sides effects of sedation during gastroscopy in healthy patients (ASA 1 and 2 patients).

Prior to propofol sedation, participants will receive either an intravenous bolus of linisol (1.5 mg/kg) = treated group or placebo = control group.

After the gastroscopy, patients will be asked to complete a satisfaction questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for gastroscopy under narcosis and who have signed the consent.
* ASA score: 1 and 2
* BMI between 18 and 30 kg/m2

Exclusion Criteria:

* Lidocaine allergy
* Anesthesia within the last 7 days
* Use of local anesthesia in the last 24 hours
* Rhythm disorder or HR <50
* Pregnant women and breastfeeding
* Participation in another clinical study in the last months
* Cannot understand VAS score or French
* Severe central nervous disease and mental illness.
* obstructive sleep apnea (known or STOP BANG score >5)
* Upper lung infection.
* Liver or kidney function disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
total propofol dose in milligramme | procedure (from the beginning of propofol infusion until arrival of the gastroscope in the stomach)
  total propofol dose consumed
total propofol dose in milligramme | Procedure (from the beginning of propofol infusion until endoscope removal)
  total propofol dose consumed
propofol in site effet concentration in microgram per milliliter | procedure (from the beginning of propofol infusion until arrival of the gastroscope in the stomach)
  AIVOC : Effect concentration of propofol
propofol in site effet concentration in microgram per milliliter | Procedure (from the beginning of propofol infusion until endoscope removal)
  AIVOC : Effect concentration of propofol

SECONDARY OUTCOMES:
number of participants with moderate hypoxemia | Procedure (during propofol sedation and gastroscopy)
  pulse saturation below 95%
number of participants with hypotension | Procedure (during propofol sedation and gastroscopy)
  mean arterial pressure below 65 mmHg
number of participants with severe hypoxemia | Procedure (during propofol sedation and gastroscopy)
  pulse saturation below 90%
number of participants presenting cough | Procedure (during propofol sedation and gastroscopy)
  cough suggesting to light sedation
number of participants presenting laryngospasm | Procedure (during propofol sedation and gastroscopy)
  laryngospasm suggesting to light sedation
number of participants presenting involuntary movements | Procedure (during propofol sedation and gastroscopy)
  involuntary movements suggesting to light sedation
number of participants presenting side effects of lidocaine administration | during gastroscopy procedure
  metallic taste, tinnitus, anaphylaxis
score of Endoscopist satisfaction (1-5) | completed procedure (before transfer to recovery room)
  Endoscopist satisfaction :1 = very bad; 2=bas; 3=good; 4=very good; 5= excellent
score of Patient satisfaction (1-5) | at recovery room discharge, an average of 1 hour after completed procedure
  Patient satisfaction :1 = very bad; 2=bas; 3=good; 4=very good; 5= excellent
throat pain | at recovery room discharge, an average of 1 hour after completed procedure
  analog digital scale from 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: celine Boudart, MD PhD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Qi XR, Sun JY, An LX, Zhang K, Xue FS. Effects of intravenous lidocaine on hypoxemia induced by propofol-based sedation for gastrointestinal endoscopy procedures: study protocol for a prospective, randomized, controlled trial. Trials. 2022 Sep 24;23(1):800. doi: 10.1186/s13063-022-06719-6. PMID 36153625
- [Background] Qi XR, Sun JY, An LX, Zhang K. Effect of intravenous lidocaine on the ED50 of propofol for inserting gastroscope without body movement in adult patients: a randomized, controlled study. BMC Anesthesiol. 2022 Oct 17;22(1):319. doi: 10.1186/s12871-022-01861-9. PMID 36253717
- [Background] Hu S, Wang M, Li S, Zhou W, Zhang Y, Shi H, Ye P, Sun J, Liu F, Zhang W, Zheng L, Hou Q, Wang Y, Sun W, Chen Y, Lu Z, Ji Z, Liao L, Lv X, Wang Y, Wang X, Yang H. Intravenous Lidocaine Significantly Reduces the Propofol Dose in Elderly Patients Undergoing Gastroscopy: A Randomized Controlled Trial. Drug Des Devel Ther. 2022 Aug 12;16:2695-2705. doi: 10.2147/DDDT.S377237. eCollection 2022. PMID 35983429